CLINICAL TRIAL: NCT00973011
Title: A Phase Ia, Multicenter, Open-Label, Single-Dose, Dose-Escalation Study of the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of Intravitreal Injections of FCFD4514S in Patients With Geographic Atrophy
Brief Title: A Study of the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of Intravitreal Injections of FCFD4514S in Patients With Geographic Atrophy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFD4711g
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Geographic Atrophy
Keywords: GA
MeSH Terms: conditions — Geographic Atrophy

ARMS (1):
- A (Experimental)
  Interventions: Drug: FCFD4514S

INTERVENTIONS:
Drug: FCFD4514S — Intravitreal escalating dose

SUMMARY:
The Phase Ia, open-label, multicenter study will consist of a single-dose, dose-escalation study of the safety, tolerability, pharmacokinetics, and immunogenicity of an intravitreal (ITV) injection of FCFD4514S in patients with Geographic Atrophy (GA).

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to undertake all scheduled visits and assessments
* Agreement to use an effective form of contraception for the duration of the study
* Geographic atrophy (GA) at least 0.75 disc areas in the absence of choroidal neovascularization (CNV)

Exclusion Criteria:

* Treatment for active systemic infection
* Predisposition or history of increased risk for infection
* Active malignancy
* History of medical conditions, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use an investigational drug or that might affect interpretation of the results of the study or that renders the patient at high risk for treatment complications
* GA in either eye due to non-AMD causes
* Active or history of ocular and intraocular conditions in the study eye (except GA)
* History of vitreoretinal surgery or laser photocoagulation in the study eye
* Prior treatment for AMD (except vitamins and minerals)
* History of intravitreal (ITV) drug delivery
* Intraocular surgery (including cataract surgery) in the study eye within 3 months preceding Day 0
* Previous participation in any studies of investigational drugs within 1 month preceding Day 0 (excluding vitamins and minerals)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of the study drug | Through study completion or early study discontinuation

SECONDARY OUTCOMES:
PK parameters of study drug (total exposure, maximum observed serum concentration, and time of maximum observed serum concentration) | Through study completion or early study discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Erich Strauss, M.D., Study Director — Genentech, Inc.